CLINICAL TRIAL: NCT02656732
Title: Clinical Evaluation of Amnion Chorion Membrane in Comparison to Subepithelial Connective Tissue Graft in Gingival Recession Coverage: A Randomized Controlled Clinical Trial.
Brief Title: Amnion Chorion Membrane in Comparison to Subepithelial Connective Tissue Graft in Gingival Recession Coverage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Noha Ayman Ghallab, Associate Professor of Oral Medicine and Periodontology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AC_SCTG
Record Dates: First submitted 2016-01-13; First posted 2016-01-15 (Estimated); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- coronally advanced flap with amnion chorion membrane (Experimental): coronally advanced flap was reflected and amnion chorion allograft membrane was placed under the flap as a guided tissue regeneration barrier.
  Interventions: Biological: amnion chorion allograft membrane
- subepithelial connective tissue graft (Active Comparator): coronally advanced flap was reflected and subepithelial connective tissue graft was harvested from the palate and placed under the flap.
  Interventions: Procedure: coronally advanced flap with the subepithelial connective tissue graft

INTERVENTIONS:
Biological: amnion chorion allograft membrane — Biologic Amnion chorion allograft membrane derived from placenta of a donor pregnant subject.
  Other Names: BioXclude™,Snoasis Medical products, USA.
  Arms: coronally advanced flap with amnion chorion membrane
Procedure: coronally advanced flap with the subepithelial connective tissue graft — coronally advanced flap with the placement of subepithelial connective tissue graft harvested from the palate
  Other Names: autogenous connective tissue graft
  Arms: subepithelial connective tissue graft

SUMMARY:
The present randomized, controlled, parallel-grouped trial included twenty patients (aged 20 to 54 years) suffering from Miller's class I or II gingival recession. Patients were randomly assigned into two equal groups; control group; the coronally advanced flap with the subepithelial connective tissue graft (CAF+SCTG) or the test group; coronally advanced flap with amnion chorion allograft membrane (CAF+AC).

DETAILED DESCRIPTION:
The participants were randomly assigned to receive coronally advanced flap (CAF) with amnion chorion membrane or CAF with subepithelial connective tissue graft using a simple randomization procedure with a 1:1 allocation ratio. A computer generated randomization list was drawn up by a faculty member who was not involved in the recruitment. Allocation concealment was achieved by sealed coded opaque envelopes that contained the treatment to be performed to the enrolled subjects based on the randomized numbers. Consequently, patients were allocated to either AC membrane (intervention) or SCTG (control) groups. The sealed envelope containing treatment assignment was opened at time of the surgery and the number was picked by another person other than the operator.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged between 18 - 60 years old.
* Subjects with facial gingival recession defects in anterior and premolar teeth classified as either class I or II defects according to Miller's classification.
* Subjects able to tolerate surgical periodontal procedures.
* Accepts the 6 months follow-up period.

Exclusion Criteria:

* Current and former smokers.
* Pregnant females.
* Subjects received any periodontal therapy for a minimum of 6 months prior to the study.
* Subjects taking drugs known to interfere with wound healing.
* Subjects with unacceptable oral hygiene with plaque index >2.
* Teeth with non-carious cervical lesions, cervical caries and malalignment.

Ages: 20 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-06; Primary Completion 2015-04 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
recession depth | Change in mm from baseline before surgical procedure to follow up at 6 months.
  It is measured as the distance from the cemento-enamel junction to the gingival margin representing the amount of root coverage.

SECONDARY OUTCOMES:
Recession Width | Change in mm from baseline before surgical procedure to follow up at 6 months.
  It is measured as the distance from mesial and distal papillae along cemento-enamel junction.
Width of keratinized gingiva | Change in mm from baseline before surgical procedure to follow up at 6 months.
  It is measured from the mucogingival junction to the free gingival margin.
Probing pocket depth | Change in mm from baseline before surgical procedure to follow up at 6 months.
  It is measuring the distance from the base of pocket to the gingival margin.
Clinical attachment level | Change in mm from baseline before surgical procedure to follow up at 6 months.
  It is measuring the distance from the apical end of periodontal probe to cemento-enamel junction.
Tissue Biotype | Change in mm from baseline before surgical procedure to follow up at 6 months.
  It is measured by penetrating the gingiva with the periodontal probe down to bone after giving local anesthesia to measure the thickness of gingival tissues
root coverage esthetic score | score taken after completion of the study at 6 months
  The clinical esthetic evaluation was performed without magnification to evaluate gingival margin, marginal tissue contour, soft tissue texture, mucogingival junction alignment and gingival color
Patient reported outcomes | taken after completion of the study at 6 months
  Patients were given certain questions regarding not regretting to perform the surgery, root hypersensitivity and aesthetic satisfaction to be answered at the 6 month follow-up for assessing their satisfaction with the whole procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Mona Shoeib, MD, Study Chair — Professor of Oral Medicine and Periodontology, Faculty of Oral and Dental Medicine, Cairo University.; Hani El-Nahas, MD, Study Director — Associate Professor of Oral Medicine and Periodontology, Faculty of Oral and Dental Medicine, Cairo University.; Manar El-Zanaty, Msc., Principal Investigator — manarzanaty@hotmail.com

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cairo F, Cortellini P, Tonetti M, Nieri M, Mervelt J, Cincinelli S, Pini-Prato G. Coronally advanced flap with and without connective tissue graft for the treatment of single maxillary gingival recession with loss of inter-dental attachment. A randomized controlled clinical trial. J Clin Periodontol. 2012 Aug;39(8):760-8. doi: 10.1111/j.1600-051X.2012.01903.x. Epub 2012 May 28. PMID 22639845
- [Result] Cairo F, Nieri M, Pagliaro U. Efficacy of periodontal plastic surgery procedures in the treatment of localized facial gingival recessions. A systematic review. J Clin Periodontol. 2014 Apr;41 Suppl 15:S44-62. doi: 10.1111/jcpe.12182. PMID 24641000
- [Result] Chambrone L, Tatakis DN. Periodontal soft tissue root coverage procedures: a systematic review from the AAP Regeneration Workshop. J Periodontol. 2015 Feb;86(2 Suppl):S8-51. doi: 10.1902/jop.2015.130674. PMID 25644302
- [Result] Chakraborthy S, Sambashivaiah S, Kulal R, Bilchodmath S. Amnion and Chorion Allografts in Combination with Coronally Advanced Flap in the Treatment of Gingival Recession: A Clinical Study. J Clin Diagn Res. 2015 Sep;9(9):ZC98-ZC101. doi: 10.7860/JCDR/2015/12971.6572. Epub 2015 Sep 1. PMID 26501023
- [Result] de Sanctis M, Zucchelli G. Coronally advanced flap: a modified surgical approach for isolated recession-type defects: three-year results. J Clin Periodontol. 2007 Mar;34(3):262-8. doi: 10.1111/j.1600-051X.2006.01039.x. PMID 17309597
- [Result] Ghahroudi AA, Khorsand A, Rokn AR, Sabounchi SS, Shayesteh YS, Soolari A. Comparison of amnion allograft with connective tissue graft for root coverage procedures: a double-blind, randomized, controlled clinical trial. J Int Acad Periodontol. 2013 Oct;15(4):101-12. PMID 24364174